CLINICAL TRIAL: NCT03325023
Title: Prospective, Randomized, Double - Blind, Placebo Controlled Trial of Dietary Modification in Conjunction With Probiotic Therapy on Clinical and Endocrinological Parameters as Well as Body Composition in Women With Polycystic Ovary Syndrome
Brief Title: Effect of Dietary Modifacation on Microbiota in Overweight and Obese Polycystic Ovary Syndrome Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: University of California, San Diego (Other); Sanprobi (Unknown)
Responsible Party: Principal Investigator, Beata Banaszewska, MD PhD Associate Proffesor Division of Infertility and Reproductive Endocrinology, Department of Gynecology and Obsterics, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PoznanUMS5
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: PCOS
Keywords: PCOS, microbiota, probiotic,obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: (Active Comparator): Dietary modification + Probiotic supplementation (Sanprobi Super Formula)
  Interventions: Dietary Supplement: Dietary and life style modification and probiotic Sanprobi Super Formula
- Placebo Comparator (Placebo Comparator): Dietary modification + placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary and life style modification and probiotic Sanprobi Super Formula — Sanprobi Super Formula consisting of: Bifidobacterium lactis, Lactobacillus acidophilus, Lactobacillus paracasei, Lactobacillus plantarum, Lactobacillus salivarius, Lactobacillus lactis, Fructooligosacharide, Inulin.
  Arms: Active Comparator:
Other: Placebo — Placebo
  Other Names: Dietary and life style modification and placebo
  Arms: Placebo Comparator

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy affecting women of reproductive age. The pathogenesis of PCOS is not fully understood. The intestinal microbiota are believed to be associated with the development of insulin resistance and obesity, and therefore contributing to the development of PCOS. Incresed permeability of the intestinal mucosal barier and absorbtion of lipoproteinase (LPS) from G (-) bacteria promotes chronic inflammation and may lead to insulin resistance.

Approximately 50-60% of women suffering from PCOS are obese. It is known that lifestyle modification and body mass reduction improves endocrine parameters and restores ovulatory menstrual cycles in most patients. Currently, the use of probiotics and prebiotics is playing an increasingly important role in the treatment of obesity through the modulation of intestinal microflora.

The objectives of the study are based on the following assumptions:

1. Insulin resistance and compensatory hyperinsulinemia are important aspects in the pathogenesis of PCOS and co-morbidity of cardiovascular disease.
2. Aberrations in the intestinal microflora are associated with the development of obesity and insulin resistance.
3. Dietary modification combined with probiotic supplementation improves endocrine and metabolic profiles in women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy affecting women of reproductive age. The pathogenesis of PCOS is not fully understood. The intestinal microbiota are believed to be associated with the development of insulin resistance and obesity, and therefore contributing to the development of PCOS. Incresed permeability of the intestinal mucosal barier and absorbtion of lipoproteinase (LPS) from G (-) bacteria promotes chronic inflammation and may lead to insulin resistance.

The microbiome consists of a complex community of microorganisms that live in the digestive tract. Intestinal microflora is colonized by various microorganisms, with the largest groups consisting of the Firmicutes, Bacteroides, Actinobacteria and Proteobacteria. Intestinal microflora has a beneficial effect on the host by competing with pathogenic bacteria, protecting the inegrity of the intestinal mucosal barier and stimulating the immune system. Some human gut microorganisms are involved In fermenting dietary fiber into short-chain fatty acids (SCFAs), such as acetic acid and butyric acid, which are then absorbed by the host. The most beneficial species of microbiota are Lactobacillus and Bifidobacterium.

Approximately 50-60% of women suffering from PCOS are obese. It is known that lifestyle modification and body mass reduction improves endocrine parameters and restores ovulatory menstrual cycles in most patients. Currently, the use of probiotics and prebiotics is playing an increasingly important role in the treatment of obesity through the modulation of intestinal microflora.

The objectives of the study are based on the following assumptions:

1. Insulin resistance and compensatory hyperinsulinemia are important aspects in the pathogenesis of PCOS and co-morbidity of cardiovascular disease.
2. Aberrations in the intestinal microflora are associated with the development of obesity and insulin resistance.
3. Dietary modification combined with probiotic supplementation improves endocrine and metabolic profiles in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent for participation in the clinical trial
2. Age 18 to 45 years Irregular menstruation (> 35 days) or secondary amenorrhea> 3 months

4. Hyperandrogenism (hirsutism and / or acne) and / or hyperandrogenemia (total serum testosterone> 0.5 ng / mL) 5. BMI > 25

Exclusion Criteria:

1. Ovarian cancer, adrenal gland tumor, endometrial cancer, cervical cancer, breast cancer
2. Congenital adrenal hyperplasia (17-OH-progesterone> 2.5 ng / mL)
3. Clinically diagnosed Cushing's disease, acromegaly, gigantism
4. Type I or II diabetes
5. Unexplained bleeding from the genital tract
6. Hormone treatment within the last 2 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-09-20 (Estimated); Study Completion 2018-10-20 (Estimated)

PRIMARY OUTCOMES:
Reduction of body mass and body fat percentage | 6 months
  Assessed using the Tanita MC-980 Body Composition Analyzer

SECONDARY OUTCOMES:
Decrease of testosterone levels | 6 months
Increased regularity of menstrual cycle | 6 months
Improved homeostasis of the intestinal microflora | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Infertility and Reproductive Endocrinology, Department of Gynecology and Obsterics, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chudzicka-Strugala I, Kubiak A, Banaszewska B, Wysocka E, Zwozdziak B, Siakowska M, Pawelczyk L, Duleba AJ. Six-month randomized, placebo controlled trial of synbiotic supplementation in women with polycystic ovary syndrome undergoing lifestyle modifications. Arch Gynecol Obstet. 2025 Feb;311(2):499-506. doi: 10.1007/s00404-024-07833-3. Epub 2024 Dec 5. PMID 39636391
- [Derived] Chudzicka-Strugala I, Kubiak A, Banaszewska B, Zwozdziak B, Siakowska M, Pawelczyk L, Duleba AJ. Effects of Synbiotic Supplementation and Lifestyle Modifications on Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2021 Aug 18;106(9):2566-2573. doi: 10.1210/clinem/dgab369. PMID 34050763